CLINICAL TRIAL: NCT02963675
Title: Incidence of Second Primary MAlignancies in pRostate Cancer Patients With bOne Metastases - an Observational Retrospective Cohort Study in Sweden (SMARCOS)
Brief Title: Incidence of Second Primary Malignancies in Prostate Cancer Patients With Bone Metastases - an Observational Retrospective Cohort Study in Sweden
Acronym: SMARCOS
Status: Completed | Type: Observational
Sponsor: Bayer (Industry)
Responsible Party: Sponsor
Other Study IDs: 18105
Record Dates: First submitted 2016-11-10; First posted 2016-11-15 (Estimated); Last update posted 2018-02-12 (Actual); Status verified 2018-02

CONDITIONS: Prostatic Neoplasms
MeSH Terms: conditions — Prostatic Neoplasms

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Retrospective
Oversight: Data Monitoring Committee: No

GROUPS / COHORTS (2):
- Group 1: Prostate cancer patients with bone metastases (mPC)
- Group 2: Castration-resistant prostate cancer patients with bone metastases (mCRPC)

INTERVENTIONS:
Other:  — external unexposed reference group

SUMMARY:
This study is conducted to obtain information about prostate cancer patients with bone metastases before the end of 2013. The incidence of second primary malignancies and overall survival in patients with castration resistant prostate cancer are of particular interest. Information from this study will serve as a historical reference for the REASSURE study (Background incidence study)

DETAILED DESCRIPTION:
Prostate cancer (PC) is the most common non-cutaneous malignancy in men. Once it becomes metastatic, it poses a serious threat to the patients' quality of life and survival. The most common site of metastases is the skeletal system: Among castration-resistant prostate cancer patients bone metastases are involved in over 90% of metastatic cases.

The development of new treatments has led to improved quality of life and prolonged lifetime among castration-resistant prostate cancer patients with metastases (mCRPC). A recent randomized clinical trial indicated significant improvement in survival and quality of life among patients with bone metastases treated with alpha emitter radium-223 as compared with placebo. To further evaluate the safety profile of Radium-223 in patients with castration resistant prostate cancer with bone metastases, Radium-223 alpha Emitter Agent in non-intervention Safety Study in mCRPC popUlation for long-teRm Evaluation (the REASSURE study), an international prospective observational single-arm cohort study was implemented as a post-marking requirement requested by the U.S. Food and Drug Administration (FDA) and European Medicines Agency (EMA).

In the case that new treatments improve the length and quality of life substantially, it can be challenging to obtain an appropriate comparison group in the post-authorization phase. This study is conducted to obtain information about prostate cancer patients with bone metastases before the end of 2013. The incidence of second primary malignancies and overall survival are of particular interest. Information from this study will serve as a historical reference for the REASSURE study

ELIGIBILITY:
Inclusion Criteria:mPC population; if the following criteria are fulfilled:

A.) PC diagnosis in 1.1.1998 - 31.12.2011 B.) Bone metastases diagnosis in 1.1.1999 - 31.12.2011 mCRPC population; if the following criteria are fulfilled:

1. PC diagnosis in 1.1.1998 - 31.12.2011
2. Bone metastases diagnosis in 1.1.2007 - 31.12.2011
3. One of the following in 1.1.2006 - 31.12.2011 and before or at the same time with bone metastases diagnosis:

   1. Discontinuation of the initial chemical castration (androgen deprivation therapy, ADT), change of the agent or modality of ADT, or start of treatment for advanced PC after the primary ADT (including chemotherapy or mitoxantrone)
   2. Surgical castration and initiation of ADT treatment, chemotherapy or mitoxantrone afterwards
   3. Treatment with medication specific to either castration-resistant PC or mCRPC (cabazitaxel, enzalutamide or abiraterone).
   4. In a sensitivity analysis, also those who have had at least 6 months since the initiation of castration treatment before cohort entry date (bone metastases diagnosis) are included in the mCRPC population.

Exclusion Criteria:

* First PC diagnosis later than 2 months after the diagnosis of bone metastases, or
* Permanent residence not in Sweden or patient otherwise not contributing to the registers at least a year before the diagnosis of bone metastases (patient counted not contributing also if database existence less than a year before cohort entry), or
* Use of any radiopharmaceuticals for bone metastases (ATC code): Samarium (V10BX02), strontium (V10BX01), rhenium (V10BX03) or radium (V10XX03).

Min Age: 18 Years | Sex: Male | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Patients with PC diagnosis in 1.1.1998 - 31.12.2013 and with bone metastases diagnosis or bone-directed treatments in 1.1.1998 - 31.12.2013 will be initially included into the large study population. From this initial population, the main analyses will concentrate on the following two populations:
  * Prostate cancer patients with bone metastases (mPC), and
  * Castration-resistant prostate cancer patients with bone metastases (mCRPC)
Sampling Method: Non-Probability Sample
Enrollment: 15953 (Actual)
Dates: Start 2016-11-15 (Actual); Primary Completion 2017-03-31 (Actual); Study Completion 2017-03-31 (Actual)

PRIMARY OUTCOMES:
Incidences of Second primary malignancies that are characterized by the following ICD-10 codes: C00-C76, C81-C96, D00-D09, D37-D48. | Up to 15 years

SECONDARY OUTCOMES:
Incidences of any site-specific second primary malignancies | Up to 15 years for mPC patients and up to 7 years for mCRPC patients
  Site-specific ICD-10 code groups from the range of all neoplasm codes C00 - D48
Overall survival | Up to 15 years for mPC patients and up to 7 years for mCRPC patients
Pathologic fracture | Up to 15 years for mPC patients and up to 7 years for mCRPC patients
  ICD-10 codes: M49.5, M84.4, M90.7
Spinal cord compression | Up to 15 years for mPC patients and up to 7 years for mCRPC patients
  ICD-10 codes: M43.9, M48.5, G95.2, G95.8
Surgery to bone | Up to 15 years for mPC patients and up to 7 years for mCRPC patients
  Based on the Nordic Medico-Statistical Committee (NOMESCO) classification of surgical procedure codes (NCSP codes)
Radiation to bone | Up to 15 years for mPC patients and up to 7 years for mCRPC patients
  Based on NCSP codes

CONTACTS AND LOCATIONS:
Overall Officials: Bayer Study Director, Study Director — Bayer
Locations (1):
- Multiple Locations, Sweden